CLINICAL TRIAL: NCT05140226
Title: Feasibility of a Home-Based Cognitive-Physical Exercise Program in Chronic Obstructive Pulmonary Disease (COPD) Patients: A Pilot Randomized Controlled Trial
Brief Title: Cognitive and Physical Training in Patients With Chronic Obstructive Pulmonary Disease Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-5336
Record Dates: First submitted 2021-11-17; First posted 2021-12-01 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Cognitive Training; Physical Training; Randomized Controlled Trial; Home-based Program; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Physical Conditioning, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Physical Training (PT) (Experimental): Participants in the PT group will perform eight weeks of home-based physical exercise training.
  Interventions: Behavioral: Physical Training
- Cognitive-Physical Training (C-PT) (Experimental): Participants in the C-PT will perform eight weeks of home-based cognitive and physical training.
  Interventions: Behavioral: Physical Training; Behavioral: Cognitive-Physical Training

INTERVENTIONS:
Behavioral: Physical Training — Eight weeks of home-based physical exercise training. Aerobic training will be performed 5 times per week using a foot peddler for a minimum of 30 minutes at a moderate intensity (Borg Exertion Scale: between 4 and 6; pedaling speed: 50 RPM). Strength training will be performed 2 times per week, with 1-3 sets of 10-12 repetitions per exercise. Strength exercises will include training with resistance bands and bodyweight exercises. Participants will be instructed to reduce the intensity of their training if they reach a score of 7 on the Borg Exertion Scale, if oxygen saturation is less than 85%, or if they experience any symptoms. Exercise prescriptions will be developed and monitored by an exercise professional with weekly follow-up meetings and supported with a web application (Physiotec) that allows customizable exercise prescriptions, tracking of exercise completion, and video tutorials.
Behavioral: Cognitive-Physical Training — Eight weeks of home-based cognitive and physical training. Cognitive training sessions will be performed 5 times per week using the Brain HQ platform (Posit Science; San Francisco, CA, USA) and will have a duration of approximately 60 minutes. The cognitive training program will be tailored by using the Personal Trainer function which presents an automated sequence of exercise levels to participants based on selected exercises. Participants will have identical sessions initially, but schedules will diverge as participants progress and as the algorithm considers their individual performance history. The Personal Trainer program will be customized to the abilities of each user and will include a focus on the following domains: sustained attention, executive function, short and long-term memory, and anxiety and depression. Participants in this group will also engage in the same exercise training intervention as participants in the Physical Training group.
  Arms: Cognitive-Physical Training (C-PT)

SUMMARY:
Cognitive and physical function impairments are common in patients diagnosed with Chronic Obstructive Pulmonary Disease (COPD). Research has shown that cognitive and physical exercise training may be a beneficial strategy to improve physical and cognitive performance in COPD patients; however, interventions combining physical and cognitive training have not been evaluated in this population. The objectives of this research are i) to evaluate the feasibility of an 8-week home-based cognitive-physical training program in COPD patients; and ii) to derive preliminary estimates on intervention efficacy with cognitive-physical training on dual-task performance, physical function, activities of daily living, and health-related quality of life. Related to our research objectives, we hypothesize that i) it will be feasible to safely recruit COPD patients into a home-based cognitive physical training program with 75% adherence and high satisfaction ratings with the prescribed training; and that ii) the combination of cognitive and physical training will be superior to physical training alone for improving dual-task and cognitive performance, physical function, activities of daily living, and health-related quality of life.

DETAILED DESCRIPTION:
Prospective study of 24 patients diagnosed with moderate to severe COPD recruited from clinics at the University Health Network (Toronto, Canada) and other local community clinics. All study assessments and interventions will be performed remotely from the participants' homes. Participants will be randomly allocated to one of the following groups and stratified by sex: i) Cognitive-Physical Training (C-PT) group: home-based cognitive training (60 minutes, 5 times per week, using the BrainHQ platform) and physical training (5 days of aerobic training and 2 days of strength training per week); ii) Physical Training (PT) group: physical exercise training alone. Study participants will have weekly follow-up video calls with the study team to review training plans. Intervention feasibility will be evaluated through recruitment rate, program adherence, satisfaction, and assessment of adverse events. Efficacy of the intervention will be assessed via cognitive performance tests (BrainHQ), dual-task performance test (i.e., spelling backwards while peddling), physical fitness assessments (i.e., lower body strength, aerobic endurance, and physical function), physical activity levels (i.e., Fitbit, physical activity questionnaire), self-reported measures of dyspnea, health-related quality of life, activities of daily living, exercise self-efficacy, and mood. Participants will have repeat assessments after 4 and 8 weeks.

Training to improve cognitive performance has shown to be successful in adults with different neurologic conditions, but has not been evaluated in COPD. The assessment of feasibility and effect estimates of home-based cognitive-physical training will serve as an important catalyst in the development of future clinical trials aimed at reducing the morbidity associated with cognitive and physical impairments in COPD.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants (≥ 50 years of age)
* Clinical and spirometric diagnosis of COPD (FEV1 30-80%)
* Access to reliable internet connection
* Ability to mobilize independently and safely, with or without a walking aid

Exclusion Criteria:

* Current participation in a pulmonary rehabilitation program
* Disease exacerbation in the past 3 months
* Diagnosis of a neurological or musculoskeletal condition that would interfere with safe performance of study tests (e.g., stroke, myopathy, inflammatory arthritis)
* Severe cognitive impairment ascertained by chart review or self-reported
* Coronary artery disease, pacemaker or implantable defibrillator, clinical diagnosis of congestive heart failure (CHF), or poorly controlled arrhythmias
* Medical instability (hepatic dysfunction, metabolic abnormalities, or active infection)
* Overt psychiatric disorder or substance abuse
* Patient on home oxygen therapy
* Insufficient English fluency and cognition to carry out testing and training
* Patient actively listed for lung transplantation

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2025-09-22 (Actual); Study Completion 2025-09-22 (Actual)

PRIMARY OUTCOMES:
Study Recruitment | Over the study period (8 weeks)
  Recruitment-success percentage and reasons for participation/non-participation in the study will be collected. A consent rate of 30% or greater has been established as our criteria to determine study feasibility for future projects.
Participant Retention in the Study | Over the study period (8 weeks)
  Participant retention will be assessed by measuring participant follow-up with testing throughout the study period. A retention rate of 80% or greater (in each group) has been established as our criteria to determine study feasibility.
Adherence to Physical Training | Over the intervention period (8 weeks)
  Adherence to the exercise training intervention will be expressed as the percentage of physical exercise activities/training days completed out of the total number of activities/training days prescribed. Adherence to the exercise intervention of 75% or greater has been established as our criteria to determine feasibility for future projects.
Adherence to Cognitive Training | Over the intervention period (8 weeks)
  Adherence to the cognitive training intervention will be expressed as i) the number of cognitive training days completed out of the total number of cognitive training days prescribed, and ii) the number of cognitive training levels and minutes completed out of the number of levels and minutes prescribed using the Brain HQ platform. Adherence to the cognitive training of 75% or greater has been established as our criteria to determine study feasibility.
Safety and Tolerability of Cognitive and Physical Training | Over the intervention period (8 weeks)
  Any adverse events with physical training will be assessed throughout the study period.
Participant Satisfaction with the Cognitive and Physical Training Interventions | Change from baseline at weeks 1, 4 and 8
  A multiple-choice and free-form questionnaire assessing the participants' satisfaction with the cognitive and physical training programs will be completed by study participants.

SECONDARY OUTCOMES:
Cognitive Function | Baseline
  The Montreal Cognitive Assessment (MoCA) will be used to screen for cognitive impairment, specifically short-term memory, visuospatial abilities, executive functions, attention, concentration, working memory, language, and orientation to time and place. The MoCA will be administered at the baseline assessment only to help characterize our study population and it takes around 10 minutes to be completed.
Physical Activity Levels | Baseline
  The International Physical Activity Questionnaire - Short Form (IPAQ-SF) will be used to measure physical activity levels in study participants. The questionnaire consists of seven questions to capture average daily time spent sitting, walking, and engaging in moderate and vigorous physical activity over the last seven days. The IPAQ-SF provides an overall physical activity level of participants based on their Metabolic Equivalent Task minutes (MET-min) per week.
Demographics Information | Baseline
  A demographic questionnaire will be administered to collect information on age, sex, ethnicity, employment status, education level, and smoking history.
Dual Task Performance | Change from baseline at 4 and 8 weeks
  Study participants will be asked to complete two single tasks and a dual-task: i) spelling backwards: spelling five letter words backwards from a list of 100 words for one minute; ii) motor task: pedaling on a foot peddler for 1 minute at a set speed of 50 RPM and at a self-selected resistance that will allow participants to hold a conversation; iii) dual-task: pedaling for 1 minute at a speed targeting 50 RPM while spelling five letter words backwards from a list of 100 words.
Cognitive Performance | Change from baseline at 4 and 8 weeks
  Participants will have their progress evaluated with cognitive training using the BrainHQ platform. BrainHQ assessments measure how the participants' performance changes and evaluate the success of the cognitive training program. Testing assignments will be personalized by using the Personal Trainer option and will have a focus on evaluating sustained attention, executive function, short and long-term memory, and anxiety and depression.
Physical Function | Change from baseline at 4 and 8 weeks
  The short physical performance battery (SPPB) will be used to assess balance, gait, lower extremity strength, and endurance. This assessment evaluates the participants' ability to stand with their feet together in several positions (side-by-side, semi-tandem, and tandem), walking speed over 4 meters, and chair stands (time to rise from a chair and return to the seated position five times).
Aerobic Endurance | Change from baseline at 4 and 8 weeks
  Aerobic endurance will be measured via a foot peddler test developed by our research group. Participants will be instructed to sit on a standard chair and to pedal at a self-selected speed for 2 minutes. After warming up, participants will continue pedaling at 50 revolutions per minute at a Borg Exertion intensity of 4. Participants will be instructed to continue pedaling for as long as they are able to maintain the current exertional intensity.
Severity of Dyspnea | Change from baseline at 4 and 8 weeks
  The Medical Research Council (MRC) Dyspnea Scale (scores 1 to 5) will be used to assess the effect of breathlessness on daily activities.
Exertional Dyspnea and Leg Fatigue | Change from baseline at 4 and 8 weeks
  The highest score on a 10-point Borg Dyspnea scale at the start and end of the Aerobic Endurance (foot peddler) test will be the primary dyspnea and leg fatigue measure.
Qualitative Descriptors of Dyspnea | Change from baseline at 4 and 8 weeks
  The 18-point Qualitative Dyspnea Scale will be ascertained at baseline and at the end of the Aerobic Endurance (foot peddler) test from a list of 18 descriptors.
Lower Body Strength | Change from baseline at 4 and 8 weeks
  The one-minute sit-to-stand test (1-STS) will be performed to evaluate lower body strength using a standard chair (46 cm). Participants will stand upright and without delay sit down again, repeating the procedure as many times as possible in a 1 min period. Participants will be instructed to indicate their Borg Dyspnea and Borg Leg Exertion scores before and after the test.
Physical Activity | 7-day intervals at week 1, week 4, and week 8
  Physical activity will be measured via an activity tracker (Fitbit, San Francisco, USA) which will record daily activity levels (minutes and steps) of the study participants.
Exercise Training | Daily over the intervention period (8 weeks)
  Exercise behaviours of the study participants will be collected via a self-reported exercise log. These logs will comprise of sections in which participants must describe the type of exercise, duration/repetitions, and intensity.
Disease Specific Quality of Life | Change from baseline at 4 and 8 weeks
  The St. George's Respiratory Questionnaire will be administered to measure the impact of COPD on overall health, daily life, and perceived well-being in our cohort. The questionnaire is composed of 50 items with scores ranging from 0 to 100 (higher scores indicate more limitations).
Impact of Symptoms on COPD | Change from baseline at 4 and 8 weeks
  The COPD Assessment Test (CAT) will be implemented to assess cough, production of phlegm, chest tightness, breathlessness, activity limitation, confidence, sleep, and energy. The CAT consists of eight items, each formatted as a six-point differential scale and with an overall score ranging from 0 to 40.
Limitations in Daily Activities | Change from baseline at 4 and 8 weeks
  The London Chest Activities of Daily Living Questionnaire will be administered to assess the limitations in performing activities of daily living as a consequence of dyspnea. It is composed of 4 domains: self-care, domestic activities, physical activities, and leisure.
Self-Efficacy to Exercise | Change from baseline at 4 and 8 weeks
  The Exercise Self-Regulatory Efficacy Scale (Ex-SRES) will be administered to measure exercise self-regulatory efficacy. The Ex-SRES is composed of 16 items asking participants to indicate the degree to which they are confident they could continue to exercise regularly when faced with different barriers. Participants will have to indicate their confidence level from 0% (not at all confident) to 100% (highly confident).
Mood | Change from baseline at 4 and 8 weeks
  The Depression, Anxiety and Stress Scale (DASS-21) questionnaire has 21 items to assess mood (anxiety, depression, and stress). There are three self-report scales designed to measure the emotional states of depression, anxiety and stress with each question ranging from a score of 0 (did not apply) to 3 (applied most of the time). Scores for each domain (depression, anxiety, and stress) will be categorized as follows: Normal, Mild, Moderate, Severe, and Extremely Severe.
Clinical Characteristics | Over the intervention period (8 weeks) and one year prior to study enrollment
  Clinical characteristics including forced expiratory volume in the first second (FEV1), medications (e.g., opioids, prednisone), baseline 6-minute walk distance, body mass index, airway obstruction, dyspnea, and exercise capacity (BODE) index, and exacerbation history will be ascertained from chart review.
Anthropometry | Change from baseline at 4 and 8 weeks
  Participants will be asked to provide data on their body weight if they have access to a weight scale at home. Otherwise, the values from their most recent pulmonary function testing will be abstracted.
Vitals | Change from baseline at 4 and 8 weeks
  Participants will be asked to provide data on their blood pressure if they have access to a blood pressure monitor. Oxygen saturation and heart rate will be measured via a pulse oximeter.
Health Care Utilization | Over the intervention period (8 weeks) and one year prior to study enrollment
  Information on health care utilization (i.e., exacerbations, use of steroid/antibiotics, mortality, admissions to hospital, history of falls, and emergency department visits) will be collected with a self-reported questionnaire administered to participants and through chart review.
Presence of Comorbidities | Over the intervention period (8 weeks) and one year prior to study enrollment
  The presence of comorbidities in our study participants will be ascertained using the Charlson Comorbidity Index and through chart review using a comprehensive comorbidity questionnaire developed by our team.

CONTACTS AND LOCATIONS:
Overall Officials: Dmitry Rozenberg, MD PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hung WW, Wisnivesky JP, Siu AL, Ross JS. Cognitive decline among patients with chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2009 Jul 15;180(2):134-7. doi: 10.1164/rccm.200902-0276OC. Epub 2009 May 7. PMID 19423714
- [Background] Holland AE, Mahal A, Hill CJ, Lee AL, Burge AT, Cox NS, Moore R, Nicolson C, O'Halloran P, Lahham A, Gillies R, McDonald CF. Home-based rehabilitation for COPD using minimal resources: a randomised, controlled equivalence trial. Thorax. 2017 Jan;72(1):57-65. doi: 10.1136/thoraxjnl-2016-208514. Epub 2016 Sep 26. PMID 27672116
- [Background] Behnke M, Taube C, Kirsten D, Lehnigk B, Jorres RA, Magnussen H. Home-based exercise is capable of preserving hospital-based improvements in severe chronic obstructive pulmonary disease. Respir Med. 2000 Dec;94(12):1184-91. doi: 10.1053/rmed.2000.0949. PMID 11192954
- [Background] Higbee DH, Dodd JW. Cognitive impairment in COPD: an often overlooked co-morbidity. Expert Rev Respir Med. 2021 Jan;15(1):9-11. doi: 10.1080/17476348.2020.1811090. Epub 2020 Aug 26. No abstract available. PMID 32811226
- [Background] Torres-Sanchez I, Rodriguez-Alzueta E, Cabrera-Martos I, Lopez-Torres I, Moreno-Ramirez MP, Valenza MC. Cognitive impairment in COPD: a systematic review. J Bras Pneumol. 2015 Mar-Apr;41(2):182-90. doi: 10.1590/S1806-37132015000004424. Epub 2015 Apr 18. PMID 25909154
- [Derived] Rozenberg D, Shore J, Camacho Perez E, Nourouzpour S, Ibrahim Masthan M, Santa Mina D, Campos JL, Huszti E, Green R, Khan MH, Lau A, Gold D, Stanbrook MB, Reid WD. Feasibility of a Home-Based Cognitive-Physical Exercise Program in Patients With Chronic Obstructive Pulmonary Disease: Protocol for a Feasibility and Pilot Randomized Controlled Trial. JMIR Res Protoc. 2023 Jul 12;12:e48666. doi: 10.2196/48666. PMID 37436794